CLINICAL TRIAL: NCT00687882
Title: Prospective Multi-Center Evaluation of the Duration of Therapy for Thrombosis in Children
Brief Title: Evaluation of the Duration of Therapy for Thrombosis in Children
Acronym: Kids-DOTT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00063928; 1U01HL130048-01A1 (NIH)
Record Dates: First submitted 2008-05-06; First posted 2008-06-02 (Estimated); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Venous Thrombosis
Keywords: Venous Thromboembolism; Postthrombotic Syndrome; Antithrombotic Therapy; Duration of Therapy; Children
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism; Postthrombotic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Intervention: A (Experimental): Patients with non-occlusive thrombus or resolved thrombosis at 6 weeks.
  Interventions: Other: Shortened duration (6 weeks) of anticoagulant therapy
- Intervention: B (Active Comparator): Patients with non-occlusive thrombus or resolved thrombosis at 6 weeks.
  Interventions: Other: Conventional duration (3 months) of anticoagulant therapy
- Parallel Cohort: Persistent Occlusive Thrombosis (Other): Patients with completely occlusive thrombosis at 6 weeks.
  Interventions: Other: No Intervention
- Parallel Cohort: Persistent Antiphospholipid Antibody (Other): Patients with persistent Positive Antiphospholipid Antibody at 6 weeks.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: Shortened duration (6 weeks) of anticoagulant therapy — Subjects with evidence of non-occlusive or resolved thrombus at 6 weeks time will be randomized to receive a total duration of anticoagulant therapy of 6 weeks.
  Arms: Intervention: A
Other: Conventional duration (3 months) of anticoagulant therapy — Subjects with evidence of non-occlusive or resolved thrombus at 6 weeks time will be randomized to receive a total duration of anticoagulant therapy of 3 months.
  Arms: Intervention: B
Other: No Intervention — Subjects with evidence of persistent thrombus at 6 weeks time will remain on anticoagulant therapy for 3-6 months at the discretion of their treating physician.
  Arms: Parallel Cohort: Persistent Occlusive Thrombosis
Other: No Intervention — Subjects with evidence of persistent antiphospholipid antibody at 6 weeks will remain on anticoagulant therapy for 3 months to indefinite duration, at the discretion of their treating physician.
  Arms: Parallel Cohort: Persistent Antiphospholipid Antibody

SUMMARY:
The Kids-DOTT trial is a randomized controlled clinical trial whose primary objective is to evaluate non-inferiority of shortened-duration (6 weeks) versus conventional-duration (3 months) anticoagulation in children with first-episode acute venous thrombosis. The first stage of the trial has consisted of a pilot/feasibility component, which then continues as the definitively-powered trial.

DETAILED DESCRIPTION:
Children (birth to 21 years of age, inclusive) with first-episode venous thrombosis in association with a reversible clinical trigger (key exclusions: history of cancer; severe thrombophilia state disclosed) are enrolled and prescribed anticoagulation according to the clinical standard of care and American College of Physicians (Chest journal) 2012 recommendations. At the 6 week (post-diagnosis) follow-up visit, repeat radiologic imaging is performed to determine residual thrombus burden and its degree of occlusion. In addition, those subjects with antiphospholipid antibodies (APA) disclosed at enrollment will undergo repeat APA testing.

Patients with residual occlusive thrombosis or persistent APA are excluded from randomization, and followed on parallel cohort arms (observational), with conventional anticoagulation durations. All other patients are randomized to a total anticoagulant duration of 6 weeks versus 3 months. Children are followed for primary efficacy endpoints of symptomatic recurrent venous thromboembolism (VTE) and primary safety endpoints of clinically-relevant bleeding (major plus clinically-relevant non-major, as per International Society of Thrombosis and Haemostasis Scientific and Standardization Committee [Journal of Thrombosis & Haemostasis] 2012 definitions/recommendations).

Children are followed through 2 years (with primary endpoint at 1 year). Those with deep venous thromboses affecting venous return from the limbs also undergo standardized post-thrombotic syndrome (PTS) outcome assessment using the Manco-Johnson pediatric PTS instrument.

The non-inferiority analysis uses a bivariate endpoint approach, modeling the inherent clinical trade-off between the risks of recurrent VTE and bleeding. The trial will enroll 750 children across 40 participating centers, and allows for a 25% rate of exclusion from the per-protocol population due to randomization non-eligibility (i.e. parallel cohort), withdrawal/loss to follow-up, and protocol non-adherence.

A sub-study, completed in late 2013, used investigational dalteparin in lieu of formulary low molecular weight heparin (typically enoxaparin) in those children who were clinically prescribed a low molecular weight heparin for sub-acute anticoagulation. The goal of this sub-study was to report dose-finding and outcomes data in children treated with dalteparin for VTE. Outcomes in these patients were qualitatively compared with those of patients who received enoxaparin, warfarin, or other anticoagulants for sub-acute anticoagulation. This portion of the study was an industry-sponsored investigator-initiated sub-study with an investigator-held IND. Since the closure of the sub-study, the overall Kids-DOTT study is no longer conducted under an Investigational New Drug (IND) application.

Principal aims and hypotheses:

Specific Aim #1: To evaluate the efficacy and safety of shortened-duration (6 weeks total) versus conventional-duration (3 months total) anticoagulation for first-episode, provoked, acute venous thrombosis among children in whom thrombus resolution/non-occlusion (i.e. established blood flow) is evident after the initial 6 weeks of anticoagulant therapy

Hypothesis: Among children with first-episode, provoked, acute venous thrombosis in whom thrombosis is resolved or non-occlusive at six weeks follow-up, a shortened duration of anticoagulation (total six weeks; i.e. no further therapy) is non-inferior in efficacy to the conventional duration (total three months) of anticoagulation with respect to the risk of symptomatic recurrent VTE at 1 year, and is superior in safety with respect to the risk of clinically-relevant bleeding.(The hypothesis will also be tested in secondary analysis at 2 years, using the same efficacy and safety outcomes as for the 1 year primary analysis.)

Specific Aim #2: To compare the composite efficacy of shortened-duration (6 weeks total) versus conventional-duration (3 months total) anticoagulation for first-episode, provoked, acute venous thrombosis among children in whom thrombus resolution/non-occlusion (i.e., blood flow) is evident after the initial 6 weeks of anticoagulant therapy.

Hypothesis: Among children with first-episode, provoked, acute venous thrombosis in whom thrombosis is resolved or non-occlusive at six weeks follow-up, a shortened duration of anticoagulation (total six weeks; i.e. no further therapy) is non-inferior to the conventional duration (total three months) of anticoagulation with respect to a composite efficacy endpoint comprised of the 1-year risk of symptomatic recurrent VTE or PTS. (The hypothesis will also be tested in secondary analysis at 2 years.)

Specific Aim #3: To determine whether outcomes of first-episode, provoked, acute venous thrombosis (specifically, with respect to recurrent VTE and PTS) among children treated with conventional-duration (3 months total) anticoagulation differ between those with and without thrombus resolution/non-occlusion at 6 weeks.

Hypothesis: Among children with first-episode, provoked, acute venous thrombosis treated with conventional-duration (3 months total) anticoagulation, the cumulative incidences of recurrent VTE and PTS are significantly lower among those in whom thrombus resolution/non-occlusion was, versus was not, evident after the initial 6 weeks of anticoagulant therapy.

Specific Aim #4: To establish a clinical trial-derived plasma and nucleic acids biorepository for future proteomic, genomic, and metabolomic investigations of predictors and modulators of VTE outcomes in children.

Specific Aim #5: To investigate whether duration of anticoagulation (over the range of 3 months to indefinite duration, as determined clinically in routine care) on influences the risks of symptomatic recurrent VTE and clinically-relevant bleeding among children with first-episode, provoked, acute venous thrombosis in whom persistent antiphospholipid antibody (APA) positivity is evident at 6- and 12 -weeks post-diagnosis.

Hypothesis: Among children with first-episode, provoked, acute venous thrombosis in whom persistent APA positivity is evident at 6- and 12 -weeks post-diagnosis, duration of anticoagulant therapy is not a predictor of symptomatic recurrent VTE but is directly related to the risk of clinically-relevant bleeding.

Specific Aim #6 (Exploratory Aim): To evaluate whether the effect of treatment duration on the risks of symptomatic recurrent VTE and clinically-relevant bleeding in children with first-episode, provoked, acute venous thrombosis differs substantively between subgroups defined by type of sub-acute anticoagulant therapy in real-world clinical use (all prescribed clinically, with the exception of investigational dalteparin, which was prescribed under an investigator-held IND through December 2013).

ELIGIBILITY:
Inclusion Criteria:

1. Children (birth to <21 years of age) with radiologically-confirmed acute deep venous thrombosis in the past 30 days
2. In the opinion of the investigator, the venous thrombosis was a provoked (i.e., non-spontaneous) event (e.g.: hospitalization; Central venous catheterization; infection; dehydration; surgery; trauma; immobility; use of estrogen-containing oral contraceptive pills; flare of autoimmune/rheumatologic condition).

Exclusion Criteria:

1. Prior episode of VTE
2. Malignancy that, in the opinion of the treating oncologist, is not in remission (note: remission may exist on or off anti-neoplastic therapy)
3. Systemic lupus erythematosus
4. Pulmonary embolism that is not accompanied by DVT or is more proximal than segmental branches of the pulmonary artery
5. Use of, or intent to use, thrombolytic therapy
6. Chronic anticoagulant at prophylactic dosing is being or will be administered beyond 6 months post VTE diagnosis
7. Moderate/severe anticoagulant deficiency (defined by any one of the following):

   1. protein C <20 IU/dL if patient is ≥3 months of age, or protein C below lower limit of detection if patient is <3 months of age;
   2. antithrombin <30 IU/dL if patient is ≥3 months of age, or antithrombin below lower limit of detection if patient is <3 months of age;
   3. protein S (free antigen or activity) <20 IU/dL.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 532 (Actual)
Dates: Start 2008-03; Primary Completion 2021-01-05 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Goldenberg, MD, PhD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (63):
- United States (54):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Orange County, Orange, California
  - Stanford Medicine, Palo Alto, California
  - UC Davis Children's Center, Sacramento, California
  - Rady Children's Hospital UCSD, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - George Washington University, Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Emory University / Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - Kosair Children's Hospital, Louisville, Kentucky
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Wayne State University, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Helen Devos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Glacier View, Kalispell, Montana
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Cornell University, Ithaca, New York
  - Cohen Children's Medical Center, New Hyde Park, New York
  - NewYork-Presbyterian, New York, New York
  - Golisano Children's Hospital, Rochester, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health Sciences University, Portland, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health, Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Texas Children's Hospital (Baylor), Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Virginia Health System University Hospital, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Medical College of Wisconsin, Blood Center of Wisconsin, Wauwatosa, Wisconsin
- Royal Children's Hospital, Parkville, Victoria, Australia
- Medizinishe Universitat Wien, Vienna, Austria
- Canada (4):
  - Stollery Children's Hospital, Edmonton, Alberta
  - McMaster Childrens Hospital, Hamilton, Ontario
  - SickKids, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Israel (2):
  - Hadassah Hebrew-University Hospital, Jerusalem
  - Sheba Medical Center, Tel Aviv
- Sophia Children's Hospital, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldenberg NA, Tripputi M, Crowther M, Abshire TC, DiMichele D, Manco-Johnson MJ, Hiatt WR. The "parallel-cohort RCT": Novel design aspects and application in the Kids-DOTT trial of pediatric venous thromboembolism. Contemp Clin Trials. 2010 Jan;31(1):131-3. doi: 10.1016/j.cct.2009.11.006. Epub 2009 Nov 24. PMID 19941974
- [Background] Kittelson JM, Spyropoulos AC, Halperin JL, Kessler CM, Schulman S, Steg G, Turpie AG, Cutler NR, Hiatt WR, Goldenberg NA; Antithrombotic Trials Leadership and Steering (ATLAS) Group. Balancing risk and benefit in venous thromboembolism trials: concept for a bivariate endpoint trial design and analytic approach. J Thromb Haemost. 2013 Aug;11(8):1443-8. doi: 10.1111/jth.12324. PMID 23773172
- [Background] Goldenberg NA, Abshire T, Blatchford PJ, Fenton LZ, Halperin JL, Hiatt WR, Kessler CM, Kittelson JM, Manco-Johnson MJ, Spyropoulos AC, Steg PG, Stence NV, Turpie AG, Schulman S; Kids-DOTT Trial Investigators. Multicenter randomized controlled trial on Duration of Therapy for Thrombosis in Children and Young Adults (the Kids-DOTT trial): pilot/feasibility phase findings. J Thromb Haemost. 2015 Sep;13(9):1597-605. doi: 10.1111/jth.13038. Epub 2015 Aug 11. PMID 26118944
- [Derived] Betensky M, Mosha M, Tarango C, Verma A, Bhat R, Kucine NE, Nakano T, Nakar C, Woods G, Amankwah E, Brandao LR, Schulman S, Goldenberg NA. Outcomes in children with provoked venous thrombosis and antiphospholipid antibodies: findings from the Kids-DOTT trial. Blood Adv. 2024 Nov 26;8(22):5790-5795. doi: 10.1182/bloodadvances.2024014415. PMID 39321425
- [Derived] Goldenberg NA, Kittelson JM, Abshire TC, Bonaca M, Casella JF, Dale RA, Halperin JL, Hamblin F, Kessler CM, Manco-Johnson MJ, Sidonio RF, Spyropoulos AC, Steg PG, Turpie AGG, Schulman S; Kids-DOTT Trial Investigators and the ATLAS Group. Effect of Anticoagulant Therapy for 6 Weeks vs 3 Months on Recurrence and Bleeding Events in Patients Younger Than 21 Years of Age With Provoked Venous Thromboembolism: The Kids-DOTT Randomized Clinical Trial. JAMA. 2022 Jan 11;327(2):129-137. doi: 10.1001/jama.2021.23182. PMID 35015038
- See also: https://www.hopkinsallchildrens.org/academics/research/multicenter-studies/kids-dott — https://www.hopkinsallchildrens.org/academics/research/multicenter-studies/kids-dott

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is as per "parallel-cohort RCT design" that certain patient subgroups specified a priori, who don't meet post-enrollment randomization criteria (randomization being at 6 weeks post-enrollment) were allocated to parallel cohort arms (observational non-randomized) for continued follow-up in the study, and for prespecified analysis separately from the RCT population.
Groups:
- Intervention: A (Shortened Duration (6 Weeks) of Anticoagulant Therapy): Patients with non-occlusive thrombus or resolved thrombosis at 6 weeks.
  Shortened duration (6 weeks) of anticoagulant therapy: Subjects with evidence of non-occlusive or resolved thrombus at 6 weeks time will be randomized to receive a total duration of anticoagulant therapy of 6 weeks.
- Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy): Patients with non-occlusive thrombus or resolved thrombosis at 6 weeks.
  Conventional duration (3 months) of anticoagulant therapy: Subjects with evidence of non-occlusive or resolved thrombus at 6 weeks time will be randomized to receive a total duration of anticoagulant therapy of 3 months.
Period: Overall Study
Arm/Group | Intervention: A (Shortened Duration (6 Weeks) of Anticoagulant Therapy) | Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy) | Parallel Cohort: Persistent Occlusive Thrombosis | Parallel Cohort: Persistent Antiphospholipid Antibody
Started | 207 | 210 | 76 | 39
Completed | 175 | 178 | 76 | 39
Not Completed | 32 | 32 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention: A (Shortened Duration (6 Weeks) of Anticoagulant Therapy) | Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy) | Parallel Cohort: Persistent Occlusive Thrombosis | Parallel Cohort: Persistent Antiphospholipid Antibody | Total
Number analyzed (Participants) | 207 | 210 | 76 | 39 | 532
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 200 | 198 | 76 | 36 | 510
  Between 18 and 65 years | 7 | 12 | 0 | 3 | 22
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (6.7) | 8.5 (6.8) | 5.6 (6.5) | 9.6 (6.9) | 8.3 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 104 | 31 | 17 | 249
  Male | 110 | 106 | 45 | 22 | 283
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: More than one race includes "other"
  Participants
    American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
    Asian | 6 | 6 | 3 | 1 | 16
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 28 | 29 | 10 | 2 | 69
    White | 151 | 146 | 57 | 31 | 385
    More than one race | 6 | 12 | 0 | 0 | 18
    Unknown or Not Reported | 16 | 16 | 5 | 5 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2 | 1 | 3 | 0 | 6
  Austria | 2 | 2 | 1 | 0 | 5
  United States | 203 | 207 | 71 | 39 | 520
  Israel | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Outcome - Occurrence of Symptomatic Recurrent Venous Thromboembolism
Description: Occurrence of symptomatic recurrent venous thromboembolism. Primary safety endpoint is occurrence of clinically-relevant bleeding (major + clinically-relevant non-major) bleeding.
Time Frame: 1 Year
Population: Per protocol population analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: A (Shortened Duration (6 Weeks) of Anticoagulant Therapy) | Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy) | Parallel Cohort: Persistent Occlusive Thrombosis | Parallel Cohort: Persistent Antiphospholipid Antibody
Number analyzed (Participants) | 154 | 143 | 76 | 39
Participants | 1 | 2 | 2 | 2

2. Primary Outcome: Safety Outcome - Occurrence of Clinically-relevant (i.e. Major Plus Clinically-relevant Non-major (CRNM)
Description: Occurrence of clinically-relevant (i.e. major plus clinically-relevant non-major (CRNM) bleeding
Time Frame: 1 year
Population: Per-protocol population used for this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: A (Shortened Duration (6 Weeks) of Anticoagulant Therapy) | Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy) | Parallel Cohort: Persistent Occlusive Thrombosis | Parallel Cohort: Persistent Antiphospholipid Antibody
Number analyzed (Participants) | 154 | 143 | 76 | 39
Participants | 1 | 1 | 2 | 2

3. Secondary Outcome: Efficacy Outcome 1 - Occurrence of Symptomatic Recurrent Venous Thromboembolism (VTE) or Development of Post Thrombotic Syndrome (PTS) (Composite Endpoint)
Description: Occurrence of symptomatic recurrent venous thromboembolism (VTE) or development of Post Thrombotic Syndrome (PTS) (composite endpoint)
Time Frame: 1 year
Population: Per protocol analysis, data not collected in the parallel cohorts.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: A ((Shortened Duration (6 Weeks) of Anticoagulant Therapy): Patients with non-occlusive thrombus or resolved thrombosis at 6 weeks.
  Shortened duration (6 weeks) of anticoagulant therapy: Subjects with evidence of non-occlusive or resolved thrombus at 6 weeks time will be randomized to receive a total duration of anticoagulant therapy of 6 weeks.
Arm/Group | Intervention: A ((Shortened Duration (6 Weeks) of Anticoagulant Therapy) | Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy) | Parallel Cohort: Persistent Occlusive Thrombosis | Parallel Cohort: Persistent Antiphospholipid Antibody
Number analyzed (Participants) | 120 | 108 | 0 | 0
Participants | 36 | 32 | 0 | 0

4. Secondary Outcome: Efficacy Outcome 2 - Occurrence of Symptomatic Recurrent Venous Thromboembolism (VTE)
Description: Occurrence of symptomatic recurrent venous thromboembolism (VTE) in the intention to treat (ITT) population.
Time Frame: 2 years
Population: Outcome events for patients with symptomatic recurrent VTE in the ITT population. Per protocol analysis, data not collected in the parallel cohorts
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: A ((Shortened Duration (6 Weeks) of Anticoagulant Therapy) | Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy) | Parallel Cohort: Persistent Occlusive Thrombosis | Parallel Cohort: Persistent Antiphospholipid Antibody
Number analyzed (Participants) | 207 | 210 | 0 | 0
Participants | 3 | 5 |  |

5. Secondary Outcome: Efficacy Outcome 3 - Development of Post Thrombotic Syndrome (PTS)
Description: Development of Post Thrombotic Syndrome (PTS)
Time Frame: 1 year
Population: Per-protocol population analysis, data not collected in the parallel cohorts
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: A ((Shortened Duration (6 Weeks) of Anticoagulant Therapy) | Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy) | Parallel Cohort: Persistent Occlusive Thrombosis | Parallel Cohort: Persistent Antiphospholipid Antibody
Number analyzed (Participants) | 120 | 108 | 0 | 0
Participants | 35 | 32 | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization up to 12 weeks plus 10 days post-diagnosis
Description: Adverse Events, Serious Adverse Events and All Cause Mortality were collected from time of randomization to the end of the 12-week study window (12 weeks plus 10 days post-diagnosis). AEs were not collected on those patients who are assigned to a parallel cohort group or withdrawn prior to randomization.
Arm/Group | Intervention: A (Shortened Duration (6 Weeks) of Anticoagulant Therapy) | Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy) | Parallel Cohort: Persistent Occlusive Thrombosis | Parallel Cohort: Persistent Antiphospholipid Antibody
All-Cause Mortality (participants affected / at risk) | 4/207 | 4/210 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 11/207 | 20/210 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 54/207 | 65/210 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: A (Shortened Duration (6 Weeks) of Anticoagulant Therapy) (N=207) | Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy) (N=210) | Parallel Cohort: Persistent Occlusive Thrombosis (N=0) | Parallel Cohort: Persistent Antiphospholipid Antibody (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 | 0
Microvillous inclusion disease (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0
Haematochesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 | 0
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 | 0
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 0 | 0
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1) | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 (2) | 0 (0) | 0 | 0
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Pneumocystic joroveci pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 | 0
Gram stain positive (Investigations) | 1 (1) | 0 (0) | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 | 0
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 | 0
Abscess drainage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 | 0
Adenotonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 | 0
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 | 0
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: A (Shortened Duration (6 Weeks) of Anticoagulant Therapy) (N=207) | Intervention: B (Conventional Duration (3 Months) of Anticoagulant Therapy) (N=210) | Parallel Cohort: Persistent Occlusive Thrombosis (N=0) | Parallel Cohort: Persistent Antiphospholipid Antibody (N=0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 | 0
Splenomegaly (Cardiac disorders) | 0 (0) | 1 (2) | 0 | 0
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 | 0
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 | 0
Microvillous inclusion disease (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 | 0
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 | 0
Otorrhea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 | 0
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 | 0
Papilledema (Eye disorders) | 1 (1) | 0 (0) | 0 | 0
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 | 0
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 | 0
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 (5) | 5 (5) | 0 | 0
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 | 0
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 | 0
Fatigue (General disorders) | 0 (0) | 1 (2) | 0 | 0
Injection site hematoma (General disorders) | 0 (0) | 3 (3) | 0 | 0
Injection site pain (General disorders) | 0 (0) | 2 (3) | 0 | 0
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 | 0
Edema peripheral (General disorders) | 0 (0) | 1 (1) | 0 | 0
Pyrexia (General disorders) | 4 (4) | 7 (7) | 0 | 0
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 0 | 0
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Bronchiolitis (Infections and infestations) | 1 (1) | 1 (1) | 0 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Celluitis (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1) | 0 | 0
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Gastric infection (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Gonorrhea (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Implant site cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 3 (3) | 0 (0) | 0 | 0
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (6) | 0 | 0
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0) | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Scrotal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (2) | 0 | 0
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 | 0
Vaginitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 | 0
Viral infection (Infections and infestations) | 2 (2) | 1 (1) | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 | 0
Albumin globulin ratio increased (Investigations) | 0 (0) | 1 (1) | 0 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 1 (1) | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 | 0
Blood osmolarity decreased (Investigations) | 0 (0) | 1 (1) | 0 | 0
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 | 0
Globulins decreased (Investigations) | 0 (0) | 1 (1) | 0 | 0
Gram stain positive (Investigations) | 1 (1) | 0 (0) | 0 | 0
International normalized ratio decreased (Investigations) | 0 (0) | 1 (1) | 0 | 0
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 | 0
Mean cell volume increased (Investigations) | 0 (0) | 1 (1) | 0 | 0
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 | 0
Transaminases increased (Investigations) | 1 (1) | 1 (1) | 0 | 0
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 | 0
Hyperkaliemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (5) | 0 | 0
Weight bearing difficulty (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 | 0
Cerebral hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 | 0
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 | 0
Headache (Nervous system disorders) | 2 (2) | 4 (5) | 0 | 0
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 0 | 0
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 | 0
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 | 0
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 | 0
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 | 0
Skin hemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 | 0
Subcutaneous hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 | 0
Abscess drainage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 | 0
Adenotonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 | 0
Ileostomy closure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 | 0
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 | 0
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 | 0

LIMITATIONS AND CAVEATS:
1. Small population of patients with cancer or pulmonary embolism
2. The anticoagulant therapies prescribed were predominantly Low Molecular Weight Heparin (LMWH), vs. oral anticoagulant therapies
3. Trade-offs between recurrent VT and current relevant bleeds
4. The secondary noninferiority analyses involving chronic venous insufficiency were solely descriptive
5. Low frequency pediatric disease with limitations
6. Small number of primary and efficacy and safety events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT00687882/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT00687882/SAP_001.pdf